CLINICAL TRIAL: NCT06955338
Title: The Effect of Music Recital and Virtual Reality on Pain, Anxiety and Fear During Oral Mucositis Care in Children With Leukaemia: A Randomised Controlled Study
Brief Title: Music and VR Effects on Pain, Anxiety, and Fear During Oral Mucositis Care in Leukaemic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, SEDA ARDAHAN SEVGİLİ, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07.03.2025/2100
Record Dates: First submitted 2025-04-22; First posted 2025-05-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Pain; Fear
Keywords: leukemia; mucositis; fear; anxiety; pain; children; nursing; symptom management
MeSH Terms: conditions — Anxiety Disorders; Pain; Leukemia; Mucositis

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Oral mucositis care will be provided by the same clinic nurse in all groups in the study and this care provider will not be blinded to the intervention. The nurse will be accompanied by a researcher at this time. This person is the person who will collect the data for the scales and will not be blinded in the study. However, the person who will do the analyses of the study tests will be blinded to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1 (No Intervention)
- Group2 (Active Comparator): Relaxing Music Session
  Interventions: Procedure: Music intervention
- Group3 (Active Comparator): Short Film Session via VR (Relaxing Nature)
  Interventions: Procedure: Virtual reality

INTERVENTIONS:
Procedure: Music intervention — The music for the study will be the 'MusiCure® 9 Scandinavia' compositions specially developed by Inge Eje and Niels Eje (Gefion Records, Copenhagen, Denmark) (MusiCure, 2024). The compositions include melodies with harp, cello, strings and sounds from nature (birds, forest and night sounds) in a soft rhythm between 60-80 bpm for relaxation, based on research into the acoustic environment of hospitals and shown to have a positive effect on patients' symptoms such as pain, fear and anxiety. Two minutes after the child starts listening to the music, oral mucositis care will be started. Five minutes after the end of the procedure, the Child Anxiety Scale-Conditioning (CAS-D), Child Fear Scale and Visual Comparison Scale will be applied and the duration of the procedure will be recorded.
  Arms: Group2
Procedure: Virtual reality — In this group, children will be shown a short film with virtual reality glasses. In the study, the short film 'MusiCure® The Journey' specially developed by Inge Eje and Niels Eje (Gefion Records, Copenhagen, Denmark) will be preferred in the virtual reality group. The duration of the film is 16 minutes (MusiCure, 2024). Two minutes after the child starts watching the film, oral mucositis care will be started. Five minutes after the end of the procedure, the duration of the procedure will be recorded by applying the Child Anxiety Scale-Conditioning (CAS-D), Child Fear Scale and Visual Comparison Scale.
  Arms: Group3

SUMMARY:
Children undergoing leukaemia treatment are exposed to a wide range of chemotherapeutic agents and immunosuppressive therapies during treatment and are therefore at great risk for complications. Mucositis is one of the leading chemotherapy-related complications affecting the quality of life of the child. Although it varies according to the degree of mucositis, oral mucosal erythema, white plaques and ulcers are extremely painful and traumatising procedures for pediatric patients during mucositis care. The pain and fear they experience during the procedure may lead children to delay/not perform oral mucositis care or not allow their parents to do so. Since mucositis is a painful condition in children, it is recommended to use distracting nonpharmacological methods that can help reduce the pain and fear of children during mucositis care. In this context, the aim of this study was to determine the effects of music and virtual reality on pain, anxiety and fear during oral mucositis care in children aged 6-12 years receiving leukaemia treatment. Block randomisation (gender (F/M) and age groups (6-9/10-12) will be used to identify participants. Five minutes before the oral mucositis care procedure, all participants, regardless of group, will be assessed with the Child Anxiety Scale-Disposition (CAS-D), Child Fear Scale and Visual Analogue Scale (VAS). The study will be conducted in three groups as control group, VR group and music group. Descriptive characteristics of dependent and independent categorical variables will be given as number and percentage, numerical descriptive characteristics will be given as mean and standard deviation. In examining the relationship between dependent and independent variables, Mann Whitney-Kruskal Wallis or Student t-Anova analyses will be performed according to the result of the analysis of conformity to normal distribution. Bonferroni analysis will be used for pairwise comparisons and Covariance analysis will be used to investigate the effect of variables with children.

ELIGIBILITY:
Inclusion Criteria:

The participant child

* is between the ages of 6-12 years
* is being followed up as an inpatient in the Paediatric Haematology Clinic
* is receiving leukaemia treatment only
* has oral mucositis
* does not have a systemic infection
* willing to participate in the study
* speak Turkish and are open to communication
* has no visual and hearing problems (not using glasses or hearing aids)

Exclusion Criteria:

* Cases not fulfilling the inclusion criteria will be excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Since leukaemia is more common in boys, biological sex will be taken as the basis for this study.
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
procedural pain | Five minutes before starting the mucositis care procedure, the child's pain will be measured and baseline pain data will be collected. Pain data will be collected again immediately after the mucositis care procedure is completed.
  The difference in pain score in different groups will be recorded.
anxiety | Five minutes before starting the mucositis care procedure, the child's anxiety will be measured and baseline data will be collected. Anxiety data will be collected again immediately after the mucositis care procedure is completed.
  The difference in anxiety score in different groups will be recorded.
fear | Five minutes before starting the mucositis care procedure, the child's fear will be measured and baseline fear data will be collected. Fear data will be collected again immediately after the mucositis care procedure is completed.
  The difference in fear score in different groups will be recorded.

SECONDARY OUTCOMES:
duration of crying | After the procedure is explained to fam/child, the duration of crying will be recorded in all groups during the mucositis intervention. The recording will last till the last moment when the equipment used for care is removed from the mouth
  The study will record the differences in crying times of children in different groups.
duration of oral mucositis care | After the procedure is explained to fam/child, the duration of procedure will be recorded in all groups. The recording will last till the last moment when the equipment used for care is removed from the mouth
  The difference in processing time in different groups will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data will not be shared for ethical reasons.